CLINICAL TRIAL: NCT01224756
Title: Safety and Efficacy of Tinoridine in the Treatment of Pain and Inflammation in Patients With Acute Tonsillitis and/or Acute Pharyngitis: a Randomized, Double-blind Study Versus Placebo
Brief Title: Efficacy of Tinoridine in Treating Pain and Inflammation in Adults
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TI-NF-1001; U1111-1116-6874 (Registry Identifier: WHO)
Record Dates: First submitted 2010-10-19; First posted 2010-10-20 (Estimated); Last update posted 2012-01-12 (Estimated); Status verified 2012-01

CONDITIONS: Pain; Inflammation
Keywords: Tonsillitis; Pharyngitis; Sore Throat; Drug Therapy
MeSH Terms: conditions — Pain; Inflammation; Tonsillitis; Pharyngitis | interventions — tinoridine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tinoridine HCl 100 mg (2 capsules) TID (Experimental)
  Interventions: Drug: Tinoridine HCl
- Placebo TID (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tinoridine HCl — Tinoridine HCl 50 mg, orally, 2 capsules three times daily for up to 4 days.
  Other Names: Nonflamin
  Arms: Tinoridine HCl 100 mg (2 capsules) TID
Drug: Placebo — Tinoridine placebo-matching capsules, orally, 2 capsules three times daily for up to 4 days.
  Arms: Placebo TID

SUMMARY:
The purpose of this study is to confirm the efficacy of tinoridine hydrochloride (HCL), three times daily (TID), in the treatment of pain and inflammation in patients with acute tonsillitis and/or acute pharyngitis of nonbacterial origin versus placebo.

DETAILED DESCRIPTION:
Tonsillitis and pharyngitis are the most common upper respiratory tract infections. The signs and symptoms are sore throat, difficulty with swallowing and/or inflamed tonsils and/or pharynx. In most cases these infections are viral in origin.

Tinoridine is a nonsteroid anti-inflammatory drug with a different mechanism of action than common nonsteroidal anti-inflammatory drugs (NSAIDs), which act by inhibiting the cyclooxygenase enzyme and thereby inhibit the synthesis of prostaglandins.

The purpose of this study is to confirm the efficacy of tinoridine in the treatment of pain and inflammation in patients with acute tonsillitis and/or acute pharyngitis of nonbacterial origin versus placebo.

ELIGIBILITY:
Inclusion Criteria:

* Participants with the following signs & symptoms: sore throat, difficulty with swallowing, and inflamed of pharynx and/or tonsils.
* Onset within 2 days

Exclusion Criteria:

* Pregnant or lactating women
* Participants hypersensitive to tinoridine
* Participants with fever, peptic ulcer, serious blood abnormality, serious hepatic impairment, serious kidney impairment
* Participants with aspirin-induced asthma
* Drug or alcohol abuse
* Participants receiving analgesic antiinflammatory drug, antibiotic and/or antiviral within 2 days before entering this study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 342 (Actual)
Dates: Start 2010-11; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Pain & Inflammatory Signs & Symptoms of Acute Tonsillitis and/or Acute Pharyngitis (Sore Throat) in participants receiving tinoridine. | Baseline and Day 5.
  The change between pain and inflammatory signs and symptoms of sore throat on day 5, and sore throat at baseline. The rating scale assesses the disappearance and improvement of pain and inflammatory signs and symptoms as a whole on a 4 point scale (0=poor with no improvement; 1=fair with improvement on day 5; 2=good with improvement on day 3 and disappearance on day 5; and 3=excellent with disappearance on day 3) with a total score range from 0 to 12. Higher scores indicate less pain and inflammatory signs and symptoms.
Pain & Inflammatory Signs & Symptoms of Acute Tonsillitis and/or Acute Pharyngitis (Painful Swallowing) in participants receiving tinoridine. | Baseline and Day 5.
  The change between pain and inflammatory signs and symptoms of painful swallowing on day 5, and painful swallowing at baseline. The rating scale assesses the disappearance and improvement of pain and inflammatory signs and symptoms as a whole on a 4 point scale (0=poor with no improvement; 1=fair with improvement on day 5; 2=good with improvement on day 3 and disappearance on day 5; and 3=excellent with disappearance on day 3) with a total score range from 0 to 12. Higher scores indicate less pain and inflammatory signs and symptoms.
Pain & Inflammatory Signs & Symptoms of Acute Tonsillitis and/or Acute Pharyngitis (Inflamed Pharynx And/Or Tonsils) in participants receiving tinoridine. | Baseline and Day 5.
  The change between pain and inflammatory signs and symptoms of inflamed pharynx and/or tonsils on day 5, and inflamed pharynx and/or tonsils at baseline. The rating scale assesses the disappearance and improvement of pain and inflammatory signs and symptoms as a whole on a 4 point scale (0=poor with no improvement; 1=fair with improvement on day 5; 2=good with improvement on day 3 and disappearance on day 5; and 3=excellent with disappearance on day 3) with a total score range from 0 to 12. Higher scores indicate less pain and inflammatory signs and symptoms.

SECONDARY OUTCOMES:
Change from Baseline in Pain Intensity Measured on a 4-Point Categorical Scale. | Baseline and Day 5.
  The change between pain intensity measured on a 4-point categorical scale on day 5 and pain intensity at baseline. The rating scale assesses a pain score on a 4 point scale (0=no pain; 1=mild pain; 2=moderate pain; and 3=severe pain) with a total score range from 0 to 12. Higher scores indicate greater pain intensity.
Change from Baseline in Visual Analogue Scale for Pain Intensity. | Baseline and Day 5.
  The change between pain intensity measured on day 5 and pain intensity at baseline. Subjects marked visual scales (in millimeters) that represented no pain to unbearable pain. Lowest Value: 0 mm. Highest Value: 100 mm. The farther to the left a subject marks, the less intense pain they feel; the farther to the right, the more pain intensity they feel. Higher numbers indicate greater pain intensity.

CONTACTS AND LOCATIONS:
Overall Officials: Professor in ENT-HN, Principal Investigator — PT. Takeda Indonesia
Locations (4):
- Indonesia (4):
  - Semarang, Central Java
  - Jakarta, DKI Jakarta
  - Surabaya, East Java
  - Bandung, West Java